CLINICAL TRIAL: NCT03313167
Title: Systematic Screening for Atrial Fibrillation-potential Patients to Increase AF Detection Rate (SCAN-AF)
Brief Title: Screening for Atrial Fibrillation (AF)-Potential Patients to Increase AF Detection Rate
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-595
Record Dates: First submitted 2017-10-12; First posted 2017-10-18 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Atrial Fibrillation-potential Patients: individuals 65 years of age or older with moderate-to-high risk of stroke
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — Non-interventional

SUMMARY:
To assess the prevalence of all (prevalent and paroxysmal) undiagnosed atrial fibrillation (AF) in a Japanese population with a moderate-to-high risk of stroke

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 and one or more of the following: hypertension, prior stroke or transient ischemic attack, congestive heart failure, diabetes mellitus, and/or vascular disease

Exclusion Criteria:

* Age < 65 years, individuals with AF or a history of AF, or individuals taking anti-arrhythmic drugs

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Japanese population with a moderate-to high risk of stroke
Sampling Method: Non-Probability Sample
Enrollment: 1316 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2019-05-23 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
number of subjects screened with AF identified at Index Visit | Up to 4 weeks
number of subjects screened with AF not identified at Index Visit | Up to 4 weeks from Index Visit
  number of subjects screened who have AF not identified at their Index Visit but subsequently found to have AF confirmed by 12-lead Electrocardiogram (ECG) during the extended monitoring period

SECONDARY OUTCOMES:
number of subjects with ECG-confirmed AF detected by the Omron BP device | Day 1 to Day 14
  number of subjects with ECG-confirmed AF detected by the Omron blood pressure (BP) device during the extended monitoring period
number of subjects with ECG-confirmed AF detected by MB or HCG-801 | Day 14 to Day 28
  number of subjects with ECG-confirmed AF detected by MyBeat (MB) or Omron HeartScan 801 (HCG-801) during the extended monitoring period
number of subjects with AF identified at Index Visit who are prescribed guideline recommended anticoagulation therapy | 24 week follow up period
number of subjects with AF identified at their Index Visit who are prescribed guideline recommended anticoagulation therapy and still on the prescribed anticoagulation therapy at the end of the 24-week follow-up period | At week 24
number of subjects with Paroxysmal atrial fibrillation (PAF) identified during the extended monitoring period who are prescribed guideline-recommended anticoagulation therapy | Day 1 to Day 28
number of subjects with PAF identified during the extended monitoring period who are prescribed guideline-recommended anticoagulation therapy and still on the prescribed anticoagulation therapy at the end of the 24-week follow-up | At week 24
number of subjects with AF identified at the Index Visit who had an ischemic stroke during the 24-week follow-up period | Index Visit up to week 24
number of subjects with PAF identified during the extended monitoring period who had an ischemic stroke during the 24-week follow-up period | Day 1 up to week 24
number of subjects with AF identified at the Index Visit who bled during the 24-week follow-up period | Index Visit up to week 24
number of subjects with PAF identified during the extended monitoring period who bled during the 24-week follow-up period | Day 1 up to week 24

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Itabashi-ku, Tokyo, Japan

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm